CLINICAL TRIAL: NCT02301481
Title: A Prospective, Randomized Phase II Trial of Neoadjuvant Chemotherapy Compared With Concomitant Boost Intensity-Modulated Radiotherapy With S-1 in Locally Advanced Gastric Adenocarcinoma
Brief Title: A Randomized Phase II Trial of Neoadjuvant Chemotherapy Compared With Chemoradiotherapy in Gastric Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Jin, M.D., MD, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC2015ST-09
Record Dates: First submitted 2014-11-23; First posted 2014-11-26 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Stomach Neoplasms; Neoadjuvant Therapy; Chemoradiotherapy; Chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); titanium silicide; Surgical Procedures, Operative; Oxaliplatin; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neoadjuvant Chemoradiotherapy (NCRT) (Experimental): NCRT arm receives intensity-modulated radiotherapy with a simultaneous integrated boost (SIB-IMRT) (45.1Gy and 40.04Gy in 22 fractions) concurrently with oral S-1(40mg/m2, orally twice daily every weekday) followed by surgery and four to six cycles of SOX at the same dosage with NCT arm.
  Interventions: Radiation: SIB-IMRT; Drug: S-1; Procedure: Surgery; Drug: SOX
- Neoadjuvant Chemotherapy (NCT) (Active Comparator): NCT arm consists of neoadjuvant three cycles of SOX(S-1: 40~60mg, orally twice daily on days 1 to 14, oxaliplatin 130mg/m2 intravenously on day 1, 21 days per cycle followed by radical surgery and another postoperative three cycles of SOX.
  Interventions: Procedure: Surgery; Drug: SOX

INTERVENTIONS:
Radiation: SIB-IMRT — 45.1Gy and 40.04Gy in 22 fractions using intensity-modulated radiotherapy with a simultaneous integrated boost (SIB-IMRT) to primary tumor
  Arms: Neoadjuvant Chemoradiotherapy (NCRT)
Drug: S-1 — 40mg/m2, orally twice daily every weekday concurrently with radiotherapy treatment
  Other Names: TS-1
  Arms: Neoadjuvant Chemoradiotherapy (NCRT)
Procedure: Surgery — Surgery, preferred D2 lymphadenectomy
Drug: SOX — SOX (S-1: 40~60mg, orally twice daily on days 1 to 14, oxaliplatin 130mg/m2 intravenously on day 1, 21 days per cycle)
  Other Names: TS-1; Oxaliplatin for injection

SUMMARY:
This prospective, randomized phase II study is designed to evaluate weather neoadjuvant chemoradiotherapy is superior to neoadjuvant chemotherapy with both followed by surgery and postoperative chemotherapy for locally advanced gastric adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven locally advanced gastric adenocarcinoma in patients staged as cT3-4N0M0 or anyTN+M0
* No distant metastasis in liver,lung,bone,central nervous system(CNS),no peritoneal transplantation
* No prior abdominal or pelvic radiotherapy
* Karnofsky performance status(KPS)≥ 70, predictive life span no less than 6 months
* Patients must have normal organ and marrow function as defined below: Leukocytes: greater than or equal to 3,000 G/L; Platelets: greater than or equal to 100,000/mm3 .Hemoglobin:greater than or equal to 10g/L .Total bilirubin: within normal institutional limits; AST/ALT: less than or equal to 1.5 times the upper limit; Creatinine within normal upper limits
* Informed consent

Exclusion Criteria:

* Any prior chemotherapy or other cancer treatment prior to this protocol
* Patients with other cancer history except cervical carcinoma in situ and non-malignant melanoma skin cancer
* With any distant metastasis in liver,lung,bone,CNS,or peritoneal transplantation
* History of allergic reactions attributed to similar chemical or biologic complex to S-1 or Xeloda or Oxaliplatin
* Uncontrolled illness including, but not limited to, active infection, symptomatic heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness
* History of myocardial infarction within the past 6 months or history of ventricular arrhythmia
* History of prior radiation to the abdomen
* Pregnant or lactating females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
R0 resection rate | 2-3 months
  The surgical procedure was total or subtotal gastrectomy with recommended D2 lymphadenectomy 4-6 weeks after neoadjuvant therapy.

SECONDARY OUTCOMES:
Pathological response rate | 2-3 months
  Pathological response were classiﬁed into three grades.Grade I signiﬁes that there is little shrinkage in the tumor; only mild regression in the tumor cells is observed under themicroscope. Grade II shows gross reduction in size of the tumor and marked regression in the cancer cells microscopically, yet viable nests of cancer tissue are still visible. Grade III implies complete or almost total resolution of the tumor on exploration, and disappearance of the tumor tissue microscopically; only remnants of degenerated cancer cells can be seen (so-called ghost cancer cells).
Tumor down-staging | 2-3 months
  Down-staging was considered as any stage reduction between clinical and pathologic stage.
Postoperative complications | 2-3 months
  During hospital stay and within the first 30 days after completion of surgery.
Acute chemotherapy/Chemoradiotherapy toxicities | 6-8 months
  chemotherapy toxicities are evaluated by NCI-CTC version 4.0 and radiotherapy toxicities are graded using the RTOG/EORTC Radiation Morbidity Scoring Schema.
Distant metastasis free survival | 3 years
Locoregional recurrence free survival | 3 years
Overall survival | 3 years

OTHER OUTCOMES:
Comparison of dosimetric differences between radiation techniques | 1 year
  To compare the dosimetric differences between the volumetric-modulated arc therapy (VMAT), Tomotherapy and intensity-modulated radiotherapy (IMRT) techniques in treatment planning.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, China

REFERENCES:
- [Derived] Wang X, Zhao DB, Yang L, Chi Y, Zhao H, Jiang LM, Jiang J, Tang Y, Li N, Liu WY, Dou LZ, Zou SM, Xue LY, Ren JS, Tian YT, Che X, Guo CG, Bai XF, Sun YM, Wang SL, Song YW, Liu YP, Fang H, Li YX, Jin J. Preoperative Concurrent Chemoradiotherapy Versus Neoadjuvant Chemotherapy for Locally Advanced Gastric Cancer: Phase II Randomized Study. Front Oncol. 2022 Apr 29;12:870741. doi: 10.3389/fonc.2022.870741. eCollection 2022. PMID 35574368